CLINICAL TRIAL: NCT05449366
Title: Intraperitoneal Paclitaxel for Patients With Primary Malignant Peritoneal Mesothelioma - a Phase I/II Dose Escalation and Safety Study
Brief Title: Intraperitoneal Paclitaxel for Patients With Primary Malignant Peritoneal Mesothelioma
Acronym: INTERACT MESO
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Erasmus Medical Center (Other)
Responsible Party: Principal Investigator, E.V.E. Madsen, Principal Investigator (MD PhD), Erasmus Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NL78373.078.21; 2021-003637-11 (EudraCT Number)
Record Dates: First submitted 2022-06-22; First posted 2022-07-08 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-01

CONDITIONS: Peritoneal Malignant Mesothelioma
Keywords: Intraperitoneal chemotherapy; Paclitaxel; Systemic chemotherapy; Palliative treatment; Dose-escalation study
MeSH Terms: interventions — Paclitaxel

STUDY DESIGN:
Intervention Model Description: A prospective, open-label, single-center, phase-1/2 study with a classic three-plus-three dose escalation design.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment arm (Experimental): According to standard of care work-up for CRS-HIPEC, patients will undergo diagnostic laparoscopy to determine the feasibility of complete cytoreduction with HIPEC. In case CRS-HIPEC is not considered feasible, a peritoneal port-a-cath (PAC) system will be placed. Through this PAC, 8-16 weekly cycles of intraperitoneal chemotherapy will be administered.
  Interventions: Drug: Intraperitoneal Paclitaxel Solution (Ml)

INTERVENTIONS:
Drug: Intraperitoneal Paclitaxel Solution (Ml) — Weekly cycles of intraperitoneal paclitaxel monotherapy
  Other Names: Paclitaxel

SUMMARY:
Patients primary malignant peritoneal mesothelioma (MPM), without extra-abdominal disease, that are not eligible (or willing) to undergo cytoreductive surgery (CRS) with hyperthermic intraperitoneal chemotherapy (HIPEC) can be included in this study. Patients will be treated with intraperitoneal (IP) chemotherapy (paclitaxel) in weekly cycles. The primary aim of this study is to determine the maximum tolerable dose (MTD) of IP monotherapy with paclitaxel for patients with MPM. The secondary aims are to assess safety and feasibility of this strategy, and to study the pharmacokinetics of paclitaxel in this setting.

DETAILED DESCRIPTION:
Malignant Peritoneal Mesothelioma (MPM) is a rare, but unfortunately very aggressive cancer with a poor prognosis. Currently, the only possibly curative treatment is cytoreductive surgery (CRS) with hyperthermic intraperitoneal chemotherapy (HIPEC). However, the majority of patients are not eligible to undergo this treatment, mainly due to extensive local disease. Currently, a palliative treatment with low morbidity is not available. Overall response rates to systemic chemotherapy are low, though morbidity rates are high. Immunotherapy presents similar shortcomings, as the morbidity rate is comparable to that of systemic chemotherapy, while its benefit for MPM patients is not proven. Especially given the high morbidity rate, and the limited effectiveness of systemic treatment with either immunotherapy or chemotherapy, there is lack of treatments suitable as palliative treatment for patients with MPM. Thereby, the majority of MPM patients currently receive no anti-tumor treatment.

As MPM very rarely disseminates outside the abdominal-cavity, the use of intraperitoneal (IP) chemotherapy seems a logical and promising step. This therapy can be delivered through an IP port-a-cath (PAC), and potentially has major advantages over systemic treatment. A higher, more effective dose of chemotherapy can directly be delivered at the site of disease, while systemic uptake is limited likely resulting in fewer toxicity. In rare cases where metastases do develop, a switch can be made to systemic treatment. By first applying local treatment, most patients will be spared a toxic and often ineffective systemic therapy. Another major advantage of the suggested approach is that ascites, a common MPM-symptom that causes major morbidity, can be drained through the same PAC-system. Paclitaxel is a well-known chemotherapeutic agent and is considered extremely favorable for IP use.

The aim of this study is to determine the maximum tolerable dose (MTD) of IP monotherapy with paclitaxel for patients with MPM, and to assess safety and feasibility of this strategy. The investigators will conduct a classic three-plus-three dose escalation study with three dose Three patients are initially enrolled into a given dose cohort. If there is no dose limiting toxicity (DLT) observed in any of these patients, the trial proceeds to enroll additional patients to the next higher dose cohort. If one patient develops a DLT at a specific dose level, three additional subjects are enrolled into that same dose cohort. Development of a DLT in more than 1 patient in a specific dose cohort (≥33%) suggests that the MTD has been exceeded, and further dose escalation is not pursued. The previous dose is considered the MTD. When the MTD is found, an expansion of 3-6 more patients in that dose cohort will be performed, to achieve a total number of 9 patients treated at the MTD-level.

Patients undergo a diagnostic laparoscopy (DLS) according to standard work-up for CRS-HIPEC. If the disease is considered not resectable, a peritoneal PAC will be placed during DLS. Through this PAC intraperitoneal paclitaxel will be administered weekly (dosage according to dose-escalation schedule). The number of cycles depends on toxicity and response to the treatment. The first response evaluation is scheduled after 8 cycles. There is no limit to the number of cycles, in case of continuing response to treatment. During the first and the fourth cycle, additional blood samples and IP-fluid samples will be collected for pharmacokinetic analysis.

ELIGIBILITY:
Inclusion Criteria:

* Histological confirmed diagnosis of malignant peritoneal mesothelioma
* Patients that are not eligible (or willing) to undergo cytoreductive surgery (CRS) with hyperthermic intraperitoneal chemotherapy (HIPEC)
* Age ≥ 18 years old
* Written informed consent according to the International Conference on Harmonisation-Good Clinical Practice (ICH-GCP) and national/local regulations
* Patients must be ambulatory, i.e. World Health Organization-Eastern Cooperative Oncology Group (WHO-ECOG) performance status 0 or 1
* Ability to return to the Erasmus Medical Center for adequate follow-up as required by this protocol
* Patients must have normal organ function and adequate bone marrow reserve as assessed by the following laboratory requirements; absolute neutrophil count >1.5 * 10^9/l, platelet count >100*10^9/l and Hemoglobin >6.0mmol /l. Patients must have a Bilirubin <1½ x upper limit of normal (ULN), Serum aspartate aminotransferase (AST) and alanine aminotransferase (ALT) <2.5 x ULN

Exclusion Criteria:

* Extra-abdominal disease/metastatic disease established by preoperative CT-scan of thorax-abdomen and/or PET-scan. Imaging not older than two months at time of surgery
* Medical or psychological impediment to probable compliance with the protocol
* Serious concomitant disease or active infections
* History of auto-immune disease or organ allografts, or with active or chronic infection, including HIV and viral hepatitis
* Serious intercurrent chronic or acute illness such as pulmonary (COPD or asthma) or cardiac (NYHA class III or IV) or hepatic disease or other illness considered by the study coordinator to constitute an unwarranted high risk for participation in this study
* Pregnant or lactating women; for all women of child-bearing potential a negative urine pregnancy test will be required as well as the willingness to use adequate contraception during the study until 4 weeks after finishing treatment
* Absence of assurance of compliance with the protocol
* An organic brain syndrome or other significant psychiatric abnormality which would comprise the ability to give informed consent, and preclude participation in the full protocol and follow-up

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2022-02-01 (Actual); Primary Completion 2025-06-01 (Actual); Study Completion 2025-08-01 (Actual)

PRIMARY OUTCOMES:
The maximum tolerable dose (MTD) | Week 3 (after two completed cycles of therapy, each cycle is 1 week)
  The primary endpoint of the study is to determine the maximum tolerable dose (MTD) of intraperitoneal (IP) paclitaxel monotherapy, for patients with malignant peritoneal mesothelioma (MPM) who are not eligible to undergo CRS-HIPEC.

SECONDARY OUTCOMES:
Toxicity assessment | Week 3 (after two completed cycles of therapy, each cycle is 1 week)
  Safety determined by toxicity assessment according to CTCAE version 5.0
Feasibility determined by the number of cycles given | Week 8 (after eight completed cycles of therapy, each cycle is 1 week)
  The treatment will be considered feasible if at least 50% of patients are able to finish 75% (i.e. 6) of total planned cycles (i.e. 8)
Area Under the Curve (AUC) | At cycle 1 and 4 (each cycle is 1 week)
  The 24-hour AUC will be calculated for systemic and intraperitoneal paclitaxel by obtaining blood and intraperitoneal fluid samples during the first and fourth treatment cycle, at time points prior to infusion, at the end of peritoneal infusion as well as every hour up to patients discharge.
Maximum concentration (Cmax) | At cycle 1 and 4 (each cycle is 1 week)
  The Cmax will be calculated by obtaining blood and intraperitoneal fluid samples during the first and fourth treatment cycle, at time points prior to infusion, at the end of peritoneal infusion as well as every hour up to patients discharge.
Elimination half life (t1/2) | At cycle 1 and 4 (each cycle is 1 week)
  The t1/2 will be calculated by obtaining blood and intraperitoneal fluid samples during the first and fourth treatment cycle, at time points prior to infusion, at the end of peritoneal infusion as well as every hour up to patients discharge.

CONTACTS AND LOCATIONS:
Locations (1):
- Erasmus Medical Center, Rotterdam, South Holland, Netherlands

IPD SHARING:
Plan to Share IPD: No